CLINICAL TRIAL: NCT04050566
Title: Analysis of Anti-malarial Immunity Development in Early Life in a Prospective Birth Cohort in Agogo, Ghana
Brief Title: Malaria Birth Cohort (MBC) in Agogo, Ghana
Acronym: MBC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bernhard Nocht Institute for Tropical Medicine (Other Government)
Collaborators: Kwame Nkrumah University of Science and Technology (Other); Kumasi Centre for Collaborative Research (KCCR) (Other); Heidelberg University (Other); KEMRI-Wellcome Trust Collaborative Research Program (Other); Agogo Presbyterian Hospital (Unknown)
Responsible Party: Principal Investigator, Dr. Jürgen May, Professor, Department Head, Bernhard Nocht Institute for Tropical Medicine
Other Study IDs: PV5940
Record Dates: First submitted 2019-08-05; First posted 2019-08-08 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Malaria
Keywords: Malaria; Immunity development; Plasmodium diversity
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mothers: 900 mothers recruited during pregnancy
- Children: 900 children born to the recruited mothers

SUMMARY:
Malaria is a major health threat worldwide with an estimated 229 million cases and 409,000 deaths in 2019 (WHO, World Malaria Report 2019). Vulnerable are young children and pregnant women. The study aims to investigate immunity development against malaria with regard to parasite, human, and socioeconomic factors and possible correlations with pathology or protection in a prospective birth cohort.

DETAILED DESCRIPTION:
Malaria during pregnancy poses substantial risks for the mother and her foetus. Due to the risk of malaria during early childhood, the study addresses the high malaria morbidity and mortality in young children. Though recognised as a public health issue, it has still not been well understood how clinical immunity against malaria parasites develops, which parasite and host factors play a role in infection susceptibility, and why some infections proceed to develop severe complications while others resolve after a mild disease.

In order to identify interactions between parasite and host, a longitudinal study is performed starting with the recruitment of pregnant women. The study is conducted in Agogo in Ghana, an area with high malaria endemicity. The study design allows to analyse the neonatal immune status at birth, after potential in-utero exposure, and follows the development of immunity over the first 36 months of life. The current paradigm is that time points and frequency of infection as well as the type of variant surface antigen expressed have an impact on the cellular and humoral immune response to malaria, the development of clinical immunity, as well as the risk for future complications.

Starting point of the study is the antenatal care visit of mothers at Agogo Presbyterian Hospital (APH) during pregnancy. During recruitment, the mother will be asked to read and sign an informed consent form approved by the local ethical committee. After consent has been obtained from the mother, biological samples are taken, and a case report form is filled. An identification card with a unique code number is handed out. The first follow-up visit occurs at the birth of the child. At this time point, samples are taken from the mothers and the child. Mothers/primary caregivers are invited to observe the EPI visits offered at their nearest health post for further follow-ups. In the first year after birth, the EPI schedule includes visits at six weeks, ten weeks, 14 weeks, six months, and nine months. During these visits, questionnaires are completed and stool samples are taken. In the first six weeks after birth, the household is visited to complete a household questionnaire including housing characteristics and household assets. Additionally, a women's questionnaire is administered, which collects demographic and socioeconomic background characteristics as well as health and related behavioural data. At 12, 18, 24, and 36 months after birth, mothers/primary caregivers are encouraged to bring their children to the study hospital (APH) for a medical check-up. For the period of 36 months after birth, mothers/primary caregivers are strongly encouraged to visit the study hospital (APH) every time the child experiences a febrile illness or a history of fever in the last week during the observation period.

ELIGIBILITY:
Inclusion Criteria:

* Catchment area of the EPI (Expanded Program of Immunization) centres with good accessibility to Agogo Prespyterian Hospital (APH)
* Willingness and able to give informed consent for herself and her child

Exclusion Criteria:

* Maternal age below 18 years
* Positive HIV status of mother
* Refusal or withdrawal of informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The study recruits pregnant women at any point during their pregnancy
Study Population: Pregnant women visiting Agogo Presbyterian Hospital (APH) for their antenatal care visit and the newborn children born to these mothers
Sampling Method: Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2019-04-08 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Malaria episodes | First 36 months of life
  Frequency and severity of malaria episodes as identified by microscopy, PCR, and clinical criteria.

SECONDARY OUTCOMES:
T cell repertoire | First 36 months of life
  T cell repertoire as measured by FACS analysis

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen May, Prof, Study Director — Bernhard Nocht Institute for Tropical Medicine; John H Amuasi, Dr, Study Director — Kwame Nkrumah University of Science & Technology (KNUST); Eva Mertens, PhD, Principal Investigator — Bernhard Nocht Institute for Tropical Medicine; Nicole Struck, PhD, Principal Investigator — Bernhard Nocht Institute for Tropical Medicine; Oumou Maiga-Ascofaré, PhD, Principal Investigator — Kumasi Centre for Collaborative Research
Locations (1):
- Agogo Presbyterian Hospital, Agogo, Ghana

IPD SHARING:
Plan to Share IPD: No